CLINICAL TRIAL: NCT04861220
Title: Pre-habilitation Program for Women Indicated to Breast Cancer Surgical Treatment.
Brief Title: Surgical Pre-habilitation in Breast Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE 42627521600005274
Record Dates: First submitted 2021-04-12; First posted 2021-04-27 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-11

CONDITIONS: Breast Neoplasm
Keywords: Breast Neoplasm; Pre-habilitation
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial in women diagnosed with breast cancer who will undergo cancer treatment with a curative therapeutic proposal. Women who attend the Hospital do Câncer III / INCA for clinical screening consultation, before starting cancer treatment, will be evaluated by physiotherapy and nutrition and recruited as to the eligibility criteria for the study. Women who agree to participate will sign the Informed Consent Form and will be submitted to an initial inclusion assessment. After recruitment and definition of their initial treatment - neoadjuvant treatment or immediate surgical treatment, women will be randomly allocated to the Intervention Group (Group A - Prehabilitation Program + neoadjuvant treatment or Group B - Prehabilitation Program + immediate surgical treatment) and Control Group (Group C - Usual activities + neoadjuvant treatment or Group D - Usual activities + immediate surgical treatment).
Who Masked: Outcomes Assessor
Masking Description: The researcher by statistical analysis will be blind, as he will not be participating in the data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-habilitation group + neoadjuvant treatment (Experimental): The patients in the Pre-habilitation group + neoadjuvant treatment (Group A), will undergo neoadjuvant cancer therapy and be instructed to practice physical exercises at home 03 times a week, during neoadjuvant therapy, until the date of surgery. The pre-habilitation program (intervention) will consist of prescription of physical exercises and guidance on its importance, through a booklet and practice practice diary. The intervention group will be accompanied weekly by a call to encourage the performance of the exercises, and in case of doubts, new explanations regarding the performance of these exercises.
  Interventions: Behavioral: Physical exercise
- Prehabilitation Program + immediate surgical treatment (Experimental): The patients in the Pre-habilitation group + immediate surgical treatment (Group B), will be instructed to practice physical exercises at home 03 times a week until the date of surgery. The pre-habilitation program (intervention) will consist of prescription of physical exercises and guidance on its importance, through a booklet and practice practice diary. The intervention group will be accompanied weekly by a call to encourage the performance of the exercises, and in case of doubts, new explanations regarding the performance of these exercises.
  Interventions: Behavioral: Physical exercise
- Usual activities + neoadjuvant treatment (No Intervention): Patients allocated to this group (Group C) will not participate in the pre-habilitation program and will be instructed to continue their usual activities during the neoadjuvant cancer therapy, until the date of surgery.
- Usual activities + immediate surgical treatment (No Intervention): Patients allocated to this group (Group D) will not participate in the pre-habilitation program and will be instructed to continue their usual activities until the date of surgery.

INTERVENTIONS:
Behavioral: Physical exercise — The prescription will be divided into 3 phases:
  Warm-up: with the object of removing the body from rest and preparing it to start the activity, it consists of exercises for upper and lower limbs, 1 minute each.
  Physical exercise: Object of physical conditioning, it consists or aerobic training with walking and muscle activation through concentric contraction of the rectus abdominis in supine position, sit and get up from a chair and resistance exercises for upper members. The patient must perform 2 sets of 12 repetitions for each exercise with a 1-minute interval between the sessions.
  Stretching and relaxing: Streching the arms above the head, stretching the legs and stretching the trunk to the left and right side will be oriented. Each stretching exercise should be done for 20 seconds. The relaxation should be performed in a sitting position, eyes closed, calm and silent place, soft breathing, for 5 minutes.
  Arms: Pre-habilitation group + neoadjuvant treatment; Prehabilitation Program + immediate surgical treatment

SUMMARY:
The National Cancer Institute estimated 625 thousand new cases of cancer (excluding cases of non-melanoma skin cancer) in Brazil for each year between 2020-2022. In 2018, there were 2.1 million new cases of breast cancer in the world, being the first in the ranking of cancers in women. Practices in healthy eating and exercise can protect and / or decrease the risk of breast cancer and improve treatment results. Breast cancer treatments cause cardiovascular changes due to age-related factors, pre-existing chronic diseases and comorbidities such as obesity, smoking and dyslipidemia. Obesity is associated with the development of several types of cancer, including breast cancer. Therapies for breast cancer have a strong association with impaired cardiac function, ranging from permanent, transient cardiotoxic effects and changes in lipid metabolism. In addition to the cardiotoxic effects, the pathophysiology of cancer and treatment favor the appearance of muscle changes, such as sarcopenia. There is sufficient evidence to support that exercise improves fitness before, during and after the completion of cancer treatment. Pre-qualification in cancer treatment is an opportunity to increase physiological reserves before neoadjuvant therapies or surgery, with the intention of improving results and accelerating recovery. It can be composed of physical exercises, nutritional interventions, and psychosocial. Excess weight or depletion are factors that negatively influence surgical and cancer outcomes. In view of the evidence, the aim of this project is to evaluate the effectiveness of physical exercise in a surgical pre-habilitation program for women diagnosed with breast cancer undergoing cancer treatment with a curative therapeutic proposal at the National Cancer Institute in Rio de Janeiro. This is a randomized clinical trial, where patients will be randomly allocated to the Intervention Group and the Control Group. The patients in the intervention group will be instructed to practice physical exercises at home until the date of surgery and those in the control group will only be instructed to maintain their usual activities. All patients will be guided individually by a nutritionist with a view to a healthier nutritional status and control of comorbidities.

DETAILED DESCRIPTION:
INTRODUCTION The National Cancer Institute estimated 625 thousand new cases of cancer (excluding non-melanoma skin cancer cases) in Brazil for each year between 2020-2022, In 2018, 2.1 million new cases of breast cancer occurred in the world , equivalent to 11.6% of all estimated cancers, being the first in the ranking of cancers for females. Among the environmental and behavioral risk factors for breast cancer, alcohol consumption, excess body weight and physical inactivity, are some of the modifiable factors. Obesity, as a risk factor for breast cancer, makes many women obese when diagnosed and when starting treatment. Adhering to healthy eating and exercise can protect and / or decrease the risk of breast cancer, in addition to improving results during and after the active phase of treatment.

After the diagnosis of the disease and evaluation of its stage, the treatment can be defined as neoadjuvant or adjuvant; systemic or regional locus. Breast cancer treatments cause cardiovascular dysfunctions, which are due to age-related factors, pre-existing chronic diseases, comorbidities such as smoking, dyslipidemia and obesity, in addition to cancer treatment.Therapies for breast cancer have a strong association with impaired cardiac function, from transient and reversible changes to permanent dysfunctions, as well as changes in lipid metabolism.

The cardiotoxic effects of cancer treatments can also affect vagal activity and, thus, influence cardiac autonomic balance. In the long run, autonomic imbalance is associated with an increased risk of cardiovascular disease and mortality, and in addition, the autonomic dysfunction that is common in many types of cancer leads to an increase in sympathetic tone and a decrease in cardiac vagal tone. As a way of assessing autonomic activity and vagal response, measures of heart rate variability (HRV) have been adopted. A reduction in parasympathetic modulation and HRV indices was observed in women with breast cancer who underwent chemotherapy, radiotherapy and hormonal therapy after one year of treatment. Physical training, which already has satisfactory results in cancer patients in relation to quality of life related to health, functionality and other aspects, also showed benefits in the autonomic modulation of patients with breast cancer. In non-cancer patients, exercise interventions show improvements in the modulation of autonomic function, minimizing cardiovascular problems and reducing mortality after episodes of myocardial infarction.

In addition to the cardiotoxic effects, cancer treatment favors the appearance of muscle changes. A systematic review with 754 women with breast cancer showed sarcopenia as a risk factor for mortality in 68% of patients. Not only the pathophysiology of cancer, but also drugs used for its treatment contribute to the loss of muscle mass.

Research indicates that physical exercise can mitigate the declines induced by cancer treatment. There is sufficient evidence to support that exercise improves fitness before, during and after treatment is completed. A cardiovascular rehabilitation program based on education and behavioral counseling offers a modification of cardiac risk, increases functional capacity, ensures monitoring of the patient's functional status, improves psychosocial well-being and can reduce recurrent hospitalizations.

Home rehabilitation can be an alternative for patients with moderate cardiac risk, self-monitoring capacity and with difficulties to attend due to social or displacement reasons. Considering the profile of the user of the Unified Health System, interventions at home and in the community seem to be the best way, together with telephone contacts for questions and / or guidance.

Pre-qualification in cancer treatment is an opportunity to increase physiological reserves even before neoadjuvant therapies or surgery, with the intention of improving results and accelerating recovery. May consist of physical exercises, nutritional and psychosocial interventions.

Knowing the nutritional profile of patients is of great importance considering the negative impact of an impaired nutritional status on postoperative outcomes. Excess weight or depletion has been reported as a factor that negatively influences surgical and cancer outcomes. The identification of patients at nutritional risk and probable sarcopenia will define an early nutritional orientation through an individualized diet with a focus on improving body composition, glycemic control, since preoperative glycemic control is associated with a lower incidence of infectious complications; and management of symptoms related to cancer treatment.

Combined with treatment, behavioral counseling is effective in motivating changes in lifestyle, which are part of the modifiable risk factors for breast cancer. Thinking about the risks that accompany the diagnosis of breast cancer, a rehabilitation focused on treating current disorders and anticipating future complications are the first steps to improve the results of care and reduce costs.

GOALS Main goal To evaluate the effectiveness of physical exercise in a surgical pre-habilitation program for women diagnosed with breast cancer who underwent cancer treatment with a curative therapeutic proposal at the Cancer Hospital III of the National Cancer Institute.

Specific objectives

* Describe the sociodemographic and clinical characteristics of the study population
* Identify the rate of adherence to physical exercise and associated factors;
* To assess changes in functional and cardiopulmonary capacity, fatigue, health-related quality of life, level of physical activity, cardiac autonomic modulation and sarcopenia in women diagnosed with breast cancer, before and after surgical treatment and throughout the follow-up periods. according to the intervention group;
* Assess the nutritional status and body composition in the inclusion of patients in the study and before surgical treatment in all participating women;
* To verify the association between regular physical exercise before surgical treatment and functional and cardiopulmonary capacity, fatigue, level of physical activity, health-related quality of life, cardiac autonomic modulation and sarcopenia in comparison with the control group;
* Describe the perception of patients regarding the performance of pre-habilitation exercises;
* To evaluate the behavioral change in the practice of physical exercises after the surgical treatment of breast cancer.

SAMPLE SIZE For the calculation of the sample size, the incidence of complications (outcomes) was considered to be 10% in the intervention group and 30% in the control group, with an alpha error of 0.05, a beta error of 0.20 and a power of 80%. Based on these parameters, it will be necessary to include 62 patients in each group. However, due to the evaluation of different outcomes and the lack of data on the incidence of complications in this population, all eligible patients will be included in the study inclusion period.

LOSS CONTROL Losses related to change, lack of information and abandonment will represent a small number, as patients remain on cancer treatment for approximately 5 years at the institution. The non-recoverable losses will have data collected from the medical records to be compared with the patients who completed the follow-up.

DATA ANALYSIS The data will be analyzed by intention to treat. The descriptive analysis will be performed by measures of central tendency and dispersion (quantitative variables) and distribution of absolute and relative frequency (qualitative variables).

To assess the normal distribution of outcomes and quantitative control variables, the Kolmogorov-Smirnov test will be performed.

To assess changes between groups in the pre- and / or post-intervention stages, the mean values will be compared by the t-student test or Mann-Whitney U test (non-parametric distribution). When analyzing the pre-verus comparison after intra-group intervention, the paired t-student test will be considered. For all analyzes, p-value less than 0.05 will be considered statistically significant.

To assess the linearity between the outcome and the quantitative adjustment variables, the dispersion diagram will be performed. Quantitative independent variables that do not have a normal distribution will be categorized. To test the collinearity of the categorical independent variables, Pearson's correlation will be performed.

To assess the association between the intervention groups and the quantitative outcomes, the differences between the means will be calculated and tested by analysis of variance, considering a value of p <0.20. Multiple linear regression will be performed using the enter method (stepwise forward), considering the 95% confidence interval. Homoscedasticity and possible biases of the model will be analyzed through residual analysis and all assumptions will be observed. To identify the explanatory power of the model, the determination coefficient will be performed. The association between intervention groups and categorical outcomes will be performed by univariate analysis, using the odds ratio (OR), assuming 95% confidence intervals (95% CI). Associations with clinical and statistical significance in the univariate analysis (considering p <0, ETHICAL AND LEGAL ASPECTS This study was submitted to the Research Ethics Committee of the National Cancer Institute (CEP / INCA), under CAAE 42627521.6.0000.5274, and approved as per opinion 4.576.731. At the time of recruitment, women will be instructed on the objectives of the study and those who agree to participate will sign the Free and Informed Consent Form (ICF).

RISK AND BENEFITS Performing physical assessments will not pose any health risks to patients. The practice of unsupervised physical exercises is safe for people without any chronic health impairment, as already mentioned in the exclusion criteria. To reduce the risks, patients will be instructed on the level of effort during the practice and on signs and symptoms of decompensation, being instructed to contact the researcher, if necessary.Despite the small risk, palpitation, excessive sweating, dizziness and shortness of breath may occur when exercising at home. If this occurs, patients will be instructed to end the exercise and contact the research team.. The study population will benefit indirectly through the results, which will analyze the effectiveness of the pre-habilitation program in improving functional capacity, fatigue, health-related quality of life, level of physical activity and autonomic modulation of women undergoing treatment for breast cancer, making it possible to plan actions to control complications.The intervention group, which will perform home physical exercises according to the guidelines, will benefit from the effects of physical exercise on physical and emotional well-being. When adhering to a healthy habit, physical conditioning, mental health and health-related quality of life improve.

FINANCING This research will not impose any burden on the institution, since patients will be evaluated on the day they attend their routine consultations and other information will be collected from the physical and / or electronic medical record. The rest of the materials will be paid for by the researchers responsible.

ELIGIBILITY:
Inclusion criteria:

- have a diagnosis of breast cancer and indication for cancer treatment with a curative therapeutic proposal

Exclusion criteria:

* having a previous cancer diagnosis
* staging IV
* practitioner of physical exercise at least 90 minutes per week
* not being able to answer the questionnaires
* be unable to practice unsupervised exercises for any reason, including: dysfunctionss orthopedic, neurological, decompensated cardiorespiratory and severe renal.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in functional capacity and muscle strength - dynamometry assessment using handgrip strength | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  The handgrip strength will be assessed using the Kratos dynamometer (model ZM - manual, Brazil). During the execution of the grasping movement, the patients are positioned seated with the adducted arm parallel to the trunk, shoulder in neutral rotation and elbow flexed at 90 °. Three measurements are made, with a minimum interval of 30 seconds between them, and the highest value obtained is considered.
Changes in functional and cardiopulmonary capacity - evaluation of the 6-minute walk test | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  The six-minute walk test will be performed in a 20-meter flat corridor, with previously demarcated distances, following the recommendations of the American Thoracic Society. Monitoring of blood pressure (BP), heart rate (HR), partial oxygen saturation (SpO2) and BORG effort perception scale will be performed before, during and after the test. For the collection of HR and SpO2 the pulse oximeter G-TECH model LED (MD 300C19) will be used and for blood pressure measurement the sphygmomanometer Heidji.
Changes cardiopulmonary capacity - evaluation of the cardiac autonomic modulation through heart rate variability. | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  It will be evaluated through the collection of HRV. Data will be extracted via Polar V800.
Changes in Sarcopenia - muscle strength and performance assessment using Time Up and Go Test | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Individuals will be asked to get up from a standard chair, walk to a marker 3 meters away and return the chair, sitting down again. The time spent will be measured with a stopwatch.
Changes in Sarcopenia - muscle strength and performance assessment using SARC-F questionnaire | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  The questionnaire consists of 5 questions for the assessment of muscle strength limitations, the ability to walk, get up from a chair, up and down stairs and experiences with falls, used to assess physical performance in sarcopenia. In 2016, a change in this questionnaire was suggested, in addition to the questions, adding the calf circumference measurement.Such an evaluation will be performed by adopting the measurement of the largest perimeter (maximum measurement in the plane perpendicular to the longitudinal line of the calf) with the patient sitting with the knees and ankles flexed at an angle of ninety degrees and feet 20 cm apart from each other using an inextensible tape ( Sanny®, model TR-4010, Brazil). The measuring tape will be passed along the entire length of the calf in an adjusted manner, but without compressing the skin. The measurements will be recorded in the nearest cm.
Changes in Sarcopenia - Evaluation of the corrected arm muscle area | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  To calculate this measure, the equations proposed by Heymsfield will be used, according to gender, using in the formula the triciptal skin fold.
Changes in functional and cardiopulmonary capacity - evaluation of the 6-minute step test | Inclusion, post chemotherapy, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  The six-minute step test will be performed with a step measuring 17 cm in height, 80 cm in width and 30 cm in length, following the same recommendations of the American Thoracic Society to the six-minute walk test. The patient must go up and down the steps for 6 minutes and the evaluator must have at the end of the test the total amount of ups and downs performed. Monitoring of blood pressure (BP), heart rate (HR), partial oxygen saturation (SpO2) and BORG effort perception scale will be performed before, during and after the test. For the collection of HR and SpO2 the pulse oximeter G-TECH model LED (MD 300C19) will be used and for blood pressure measurement the sphygmomanometer Heidji.

SECONDARY OUTCOMES:
Changes in Nutritional Risk | Inclusion and pre-surgical moment
  Evaluation through the Global Subjective Assessment Produced by the Patient (ASG-PPP).
Changes in Fatigue | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Evaluation through the FACIT-Fatigue 4th version Questionnaire (Functional Assessment of Chronic Illness Therapy-Fatigue)
Changes in Physical activity level | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Evaluation through the International Physical Activity Questionnaire (IPAQ) - short version.
Changes in Health-related quality of life | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Evaluation through the EORTC QLQ-C30 3rd version
Assessment of adherence to physical exercises | pre-surgical moment
  Through the exercise diary, in which group A patients will be instructed to fill it out daily during the intervention period. In this diary, patients must inform the types of exercises performed each day, as well as the degree of difficulty and intensity.
Assessment of behavioral change in physical exercise | pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Evaluation through the International Physical Activity Questionnaire - long version.
Evaluation of the patients' perception regarding the performance of the exercises | pre-surgical moment
  For the intervention group, at the time of the post-intervention assessment, a questionnaire will be applied with 15 pre-established questions about the experience regarding the educational material received, as well as regarding the performance of the exercises. The professional who will ask the questions in this questionnaire will not be the same person who carried out the guidelines and made the weekly phone calls, so that there is no bias in the answers.
Changes in alcohol consumption and smoking | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  Evaluation through the Behavioral Risk Factor Surveillance System - BRFSS questionnaire
Changes in anthropometric data through body weight assessment | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  For the measurement of body weight, the patient will be instructed to stand up right, in the center of the scale, without shoes and wearing light clothing. You will be asked to distribute your body weight evenly over your feet. The scale used will be a portable digital type (Welmy®, model 110, Brazil), with a maximum capacity of 150 (kilogram; Kg) and accuracy of 100 (gram; g)
Evaluation of anthropometric data by height | Inclusion
  To measure the height (meter; m), a measuring tape fixed on the wall will be used. The measurement will be performed with the patient standing, barefoot or wearing thin stockings, and with as little clothing as possible so that the position of the body can be seen by the examiner. He will be instructed to stand in an orthostatic position looking at a fixed point at eye level (Frankfurt horizontal plane), to distribute the weight equally between both feet and to keep the arms freely loose along the trunk, with the palms facing the thighs.
Changes in anthropometric data through tricipital skin fold assessment | Inclusion, pre-surgical moment, 30 days after surgery, 6 months after surgery and 1 year after surgery.
  For measurement, the fatty tissue will be slightly detached from the muscle tissue and clamped with the calibrator forming a right angle exactly at the marked location. The arm should be kept relaxed and released at the side of the body during the measurement. The measurement will be determined parallel to the longitudinal axis of the dominant arm, and there may be changes with the appearance of some postoperative complication in the limb to be evaluated, on the posterior face, with the exact point of repair being the distance between the acromion and the olecranon, following the same technique described for BP measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Simone A Saraiva, Principal Investigator — Instituto Nacional de Cancer, Brazil
Locations (1):
- Instituto Nacional do Câncer / HCIII, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No